CLINICAL TRIAL: NCT00985166
Title: Administration of Frozen Measles, Mumps, Rubella, and Varicella (MMRV) Vaccine to Healthy Children at 4 to 6 Years of Age
Brief Title: A Study of ProQuad in Healthy 4 to 6 Year Old Children (V221-014)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V221-014; 2009_668
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Results first posted 2010-01-29 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): ProQuad + Placebo
  Interventions: Biological: ProQuad (Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live); Biological: Comparator: Placebo
- 2 (Active Comparator): M-M-R II + Placebo
  Interventions: Biological: Comparator: M-M-R II; Biological: Comparator: Placebo
- 3 (Active Comparator): M-M-R II + Varivax
  Interventions: Biological: Comparator: M-M-R II; Biological: Comparator: Varivax

INTERVENTIONS:
Biological: ProQuad (Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live) — A Single 0.5 mL subcutaneous injection at Day 1
  Other Names: ProQuad
  Arms: 1
Biological: Comparator: M-M-R II — A Single 0.5 mL subcutaneous injection at Day 1
  Arms: 2; 3
Biological: Comparator: Varivax — A Single 0.5 mL subcutaneous injection at Day 1
  Arms: 3
Biological: Comparator: Placebo — A Single 0.5 mL subcutaneous placebo injection at Day 1
  Arms: 1; 2

SUMMARY:
The study was conducted to determine if ProQuad may be used in place of the second dose of M-M-R II routinely given to children 4 to 6 years old who were previously immunized with M-M-R II and Varivax.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* Received primary dose of M-M-R II at less than or equal to 12 months of age
* Received primary dose of Varivax at less than or equal to 12 months of age
* Negative history of varicella, zoster, measles, mumps, and rubella

Exclusion Criteria:

* history of receiving more than once dose of M-M-R II or Varivax
* Any immune impairment or deficiency
* Exposure to measles, mumps, rubella, varicella, or zoster in the 4 weeks prior to vaccination
* Vaccination with an inactive vaccine with in the past 14 days
* Vaccination with a live vaccine within the past 30 days
* Receipt of immune globulin, or blood product in the past 5 months

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 801 (Actual)
Dates: Start 2000-08; Primary Completion 2002-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Reisinger KS, Brown ML, Xu J, Sullivan BJ, Marshall GS, Nauert B, Matson DO, Silas PE, Schodel F, Gress JO, Kuter BJ; Protocol 014 Study Group for ProQuad. A combination measles, mumps, rubella, and varicella vaccine (ProQuad) given to 4- to 6-year-old healthy children vaccinated previously with M-M-RII and Varivax. Pediatrics. 2006 Feb;117(2):265-72. doi: 10.1542/peds.2005-0092. PMID 16452343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 clinical sites in the United States
  Date of first participant visit: 24-Aug-2000
  Date of last participant visit: 06-May-2002
Pre-assignment Details: Prior to entering study, all subjects received primary dose of M-M-R II™ and Varivax™ at less than or equal to 12 months of age.
Groups:
- ProQuad™ + Placebo: ProQuad™ (measles, mumps, rubella, and varicella vaccine) + placebo administered concomitantly at separate injection sites on Day 1.
- M-M-R™ II + Placebo: M-M-R™ II + placebo administered concomitantly at separate injection sites on Day 1.
- M-M-R™ II + VARIVAX™: VARIVAX™ + M-M-R™ II administered concomitantly at separate injection sites on Day 1.
Period: Overall Study
Arm/Group | ProQuad™ + Placebo | M-M-R™ II + Placebo | M-M-R™ II + VARIVAX™
Started | 401 (Two randomized subjects withdrew consent before vaccination: no demographic information available.) | 205 | 195
Vaccinated at Visit 1 | 399 | 205 | 195
Completed | 392 | 201 | 188
Not Completed | 9 | 4 | 7
Not completed — Lost to Follow-up | 3 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 2 | 0
Not completed — Test not done | 2 | 0 | 4
Not completed — Other | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ProQuad™ + Placebo | M-M-R™ II + Placebo | M-M-R™ II + VARIVAX™ | Total
Number analyzed (Participants) | 399 | 205 | 195 | 799
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.3 (0.5) | 4.3 (0.5) | 4.3 (0.5) | 4.3 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 105 | 77 | 373
  Male | 208 | 100 | 118 | 426
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 49 | 19 | 25 | 93
  Asian/Pacific | 8 | 5 | 3 | 16
  Caucasian | 313 | 162 | 153 | 628
  Hispanic | 15 | 10 | 7 | 32
  Other | 14 | 9 | 7 | 30

OUTCOME MEASURES:

1. Primary Outcome: Antibody Response to Varicella for Subjects Who Had Previously Received M-M-R II + VARIVAX - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to Varicella
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, received M-M-R™ II + VARIVAX™ prior to entering the study, and followed protocol procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | ProQuad™ + Placebo | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 367 | 171
gpELISA units/mL | 322.2 [278.9 to 372.2] | 209.3 [171.2 to 255.9]

2. Primary Outcome: Antibody Response to Measles for Subjects Who Had Previously Received M-M-R II + VARIVAX - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to Measles
Time Frame: 6 weeks Postvaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | ProQuad™ + Placebo | M-M-R™ II + Placebo | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 367 | 185 | 171
mIU/mL | 1985.9 [1817.6 to 2169.9] | 2046.9 [1815.2 to 2308.2] | 2084.3 [1852.3 to 2345.5]

3. Primary Outcome: Antibody Response to Mumps for Subjects Who Had Previously Received M-M-R II + VARIVAX - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to Mumps
Time Frame: 6 weeks Postvaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA AB units/mL
Arm/Group | ProQuad™ + Placebo | M-M-R™ II + Placebo | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 367 | 185 | 171
ELISA AB units/mL | 206.0 [188.2 to 225.4] | 308.5 [269.6 to 352.9] | 295.9 [262.5 to 333.5]

4. Primary Outcome: Antibody Response to Rubella for Subjects Who Had Previously Received M-M-R II + VARIVAX - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to Rubella
Time Frame: 6 weeks Postvaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | ProQuad™ + Placebo | M-M-R™ II + Placebo | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 367 | 185 | 171
IU/mL | 217.3 [200.1 to 236.0] | 174.0 [157.3 to 192.6] | 154.1 [138.9 to 170.9]

ADVERSE EVENTS:
Description: The number of participants listed as "at risk" is the number of participants with follow-up.
  0/0 indicates that subjects in this treatment group did not receive the indicated vaccine.
Arm/Group | ProQuad™ + Placebo | M-M-R™ II + Placebo | M-M-R™ II + VARIVAX™
Serious Adverse Events (participants affected / at risk) | 1/397 | 0/205 | 0/193
Other Adverse Events (participants affected / at risk) | 292/397 | 150/205 | 140/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ProQuad™ + Placebo (N=397) | M-M-R™ II + Placebo (N=205) | M-M-R™ II + VARIVAX™ (N=193)
Pyelonephritis - Not other wise Specified (NOS) (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ProQuad™ + Placebo (N=397) | M-M-R™ II + Placebo (N=205) | M-M-R™ II + VARIVAX™ (N=193)
Ear pain (Ear and labyrinth disorders) | 9 | 1 | 4
Conjunctivitis (Eye disorders) | 5 | 2 | 2
Lacrimation increased (Eye disorders) | 1 | 0 | 2
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 10 | 4 | 3
Diarrhoea NOS (Gastrointestinal disorders) | 14 | 7 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 1 | 2
Vomiting NOS (Gastrointestinal disorders) | 23 | 7 | 8
Influenza like illness (General disorders) | 4 | 4 | 0
Malaise (General disorders) | 2 | 0 | 2
Pain NOS (General disorders) | 6 | 1 | 0
Pyrexia (General disorders) | 41 | 20 | 19
Venipuncture site pain (General disorders) | 0 | 2 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 2
Ear infection NOS (Infections and infestations) | 4 | 1 | 3
Gastroenteritis viral NOS (Infections and infestations) | 4 | 1 | 2
Nasopharyngitis (Infections and infestations) | 52 | 26 | 26
Otitis media NOS (Infections and infestations) | 12 | 9 | 10
Pharyngitis (Infections and infestations) | 2 | 7 | 3
Pharyngitis streptococcal (Infections and infestations) | 6 | 3 | 2
Pneumonia NOS (Infections and infestations) | 3 | 1 | 2
Sinusitis NOS (Infections and infestations) | 6 | 6 | 1
Upper respiratory tract infection NOS (Infections and infestations) | 18 | 10 | 9
Viral infection NOS (Infections and infestations) | 1 | 1 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 5 | 4 | 2
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 2
Appetite decreased NOS (Metabolism and nutrition disorders) | 4 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1
Headache (Nervous system disorders) | 22 | 10 | 12
Somnolence (Nervous system disorders) | 1 | 0 | 3
Irritability (Psychiatric disorders) | 9 | 3 | 4
Asthma NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Bronchospasm NOS (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 18 | 21
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 17 | 18 | 7
Dermatitis contact (Skin and subcutaneous tissue disorders) | 6 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 3
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Rash NOS (Skin and subcutaneous tissue disorders) | 7 | 6 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Injection site bruising (M-M-R II Injection-site) (General disorders) | 0/0 | 5 | 3
Injection site erythema (M-M-R II Injection-site) (General disorders) | 0/0 | 32 | 28
Injection site pain (M-M-R II Injection-site) (General disorders) | 0/0 | 75 | 68
Injection site swelling (M-M-R II Injection-site) (General disorders) | 0/0 | 21 | 15
Injection site bruising (ProQuad Injection-site) (General disorders) | 14 | 0/0 | 0/0
Injection site erythema (ProQuad Injection-site) (General disorders) | 98 | 0/0 | 0/0
Injection site pain (ProQuad Injection-site) (General disorders) | 163 | 0/0 | 0/0
Injection site pruritus (ProQuad Injection-site) (General disorders) | 4 | 0/0 | 0/0
Injection site rash (ProQuad Injection-site) (General disorders) | 7 | 0/0 | 0/0
Injection site swelling (ProQuad Injection-site) (General disorders) | 62 | 0/0 | 0/0
Injection site bruising (Varivax Injection-site) (General disorders) | 0/0 | 0 | 4
Injection site erythema (Varivax Injection-site) (General disorders) | 0/0 | 0 | 31
Injection site nodule (Varivax Injection-site) (General disorders) | 0/0 | 0 | 2
Injection site pain (Varivax Injection-site) (General disorders) | 0/0 | 0 | 71
Injection site pruritus (Varivax Injection-site) (General disorders) | 0/0 | 0 | 2
Injection site swelling (Varivax Injection-site) (General disorders) | 0/0 | 0 | 21

LIMITATIONS AND CAVEATS:
GMTs (adjusted for prevaccination titer, study center, and primary vaccination history status) have been reported in the literature. One subject received diluent only at visit 1 and was excluded from all immunogenicity/safety summaries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.